CLINICAL TRIAL: NCT03701048
Title: Intraoperative and Postoperative Results of Rectus Musle Reapproximation During Cesarean Section
Brief Title: Rectus Musle Reapproximation During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018/10
Record Dates: First submitted 2018-10-06; First posted 2018-10-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reappoximation of rectus muscle (Active Comparator): During Cesarean Section rectus muscle will be reapproximated with interrupted sutures.
  Interventions: Procedure: Cesarean Section
- no reappoximation of rectus muscle (Active Comparator): During Cesarean Section rectus muscle will not be closed.
  Interventions: Procedure: Cesarean Section

INTERVENTIONS:
Procedure: Cesarean Section — Pfnannenstiel incision will be done under general or spinal anaesthesia. The abdomen will be opened and fetus and plasenta will be delivered. Then abdomen will be closed.

SUMMARY:
During Cesarean section in Group 1 rectus muscle will be closed with interrupted sutures. In group 2 rectus muscle will not be closed. Postoperative pain scores, distance between the rectus muscles and bowel functions will be evaluated.

DETAILED DESCRIPTION:
Pfannenstiel incision will be done under general or spinal anesthesia. The abdomen will be opened and fetus and placenta will be delivered. Then the abdomen will be closed. In Group 1 rectus muscle will be closed with interrupted sutures. In group 2 rectus muscle will not be closed. Postoperative pain scores, distance between the rectus muscles and bowel functions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old women undergoing cesarean section

Exclusion Criteria:

* grandmultiparas

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain: Visual Analog Score | 24 hours after the procedure
  Visual Analog Scores, minimum score is 0, maximum score is 10. Score 10 represents highest pain score.
Postoperative interrectus distance | 6 weeks after the procedure
  Distance between the margins of the rectus muscles in centimeters will be measured with ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan A Çetin, Principal Investigator — KSSTRH
Locations (1):
- Kanuni SSRTH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyell DJ, Naqvi M, Wong A, Urban R, Carvalho B. Rectus Muscle Reapproximation at Cesarean Delivery and Postoperative Pain: A Randomized Controlled Trial. Surg J (N Y). 2017 Aug 11;3(3):e128-e133. doi: 10.1055/s-0037-1604074. eCollection 2017 Jul. PMID 28840194